CLINICAL TRIAL: NCT05181020
Title: Studying the Influence of Exposure to Maternal Voice on Oral Feeding Volumes in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Shabnam Lainwala, Principal Investigator, Attending Neonatologist, Connecticut Children's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-026
Record Dates: First submitted 2021-12-13; First posted 2022-01-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2023-02

CONDITIONS: Enteral Feeding
Keywords: Maternal Voice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Maternal Voice Exposure (Experimental): Infants enrolled will be exposed to maternal voice for 20 min immediately prior to being offered oral feedings. This exposure will be conducted 2 times a day until infant starts taking all enteral feeds orally.
  Interventions: Behavioral: Maternal Voice Exposure

INTERVENTIONS:
Behavioral: Maternal Voice Exposure — Main objective of this study is to determine if it is possible to expose preterm infant in a systematic manner to mother's voices before their feeds and to determine if this exposure results in an increase in their oral intake.

SUMMARY:
Oral feeding is one of the primary functions of the neonatal brain. In preterm infant population, competency at oral feeding is one of the major milestones in preparation for discharge. Mother's voices have been shown to have a net stimulatory effect and premature infants have been found to have increased cardiorespiratory stability after listening to mother's voices. Main objective of this study is to determine if it is possible to expose preterm infant in a systematic manner to mother's voices before their feeds and to determine if this exposure results in an increase in their oral intake.

DETAILED DESCRIPTION:
Achievement of full oral feedings is directly associated with length of neonatal intensive care unit stay. Extremely low gestational age infants with dysfunctional oral feeding in early childhood have lower cognitive and language skills compared with those with normal oral feedings. Also, previous studies have shown a strong association between oral feeding and infant maturity and behavior state and positive feeding experience. In recent years, there is emerging evidence that non-medical developmental care interventions in the neonatal intensive care units such as kangaroo care, single family rooms, and music and massage therapy may be beneficial for preterm infants and improve their long term neurodevelopmental outcomes. Beneficial effects of exposure to mother's voice and sounds on preterm infants in the neonatal intensive care units are well documented. Our study proposes to examine the association between exposure to mother's voice prior to and during oral feeding and oral feeding volume and rate in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between gestational age of 28 0/7 weeks and 34 6/7 weeks
* Ready to start oral feeding attempts
* Taking a total daily oral intake < 50% of feeds on average in 2 days prior to starting intervention
* Mothers who are English speaking and over 18 years old

Exclusion Criteria:

* Major congenital anomalies
* Non-English speaking
* Family history of suspected congenital hearing loss
* Failed hearing test in NICU
* Grade three to four intraventricular hemorrhage or periventricular leukomalacia
* necrotizing enterocolitis requiring treatment
* Congenital infections such as cytomegalovirus which can lead to sensorineural hearing loss

Ages: 28 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Oral feeding volume | Through study completion, average 40 weeks post menstrual age
  Effect of maternal voice immediately prior to feeding on oral feeding volumes in preterm infants

CONTACTS AND LOCATIONS:
Overall Officials: Shabnam Lainwala, MBBS, PhD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chhikara A, Hagadorn JI, Lainwala S. Effect of maternal voice on proportion of oral feeding in preterm infants. J Perinatol. 2023 Jan;43(1):68-73. doi: 10.1038/s41372-022-01493-4. Epub 2022 Aug 18. PMID 35982244